CLINICAL TRIAL: NCT05638919
Title: Real-world Effectiveness of Oral Antivirals for Treatment of COVID-19 in Ministry of Health Malaysia Institutions
Brief Title: Real World COVID-19 Antiviral Effectiveness Research
Acronym: myRECOVER
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Clinical Research Centre, Malaysia (Other)
Responsible Party: Sponsor
Other Study IDs: NMRR ID-22-00938-2YN
Record Dates: First submitted 2022-12-04; First posted 2022-12-06 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: COVID-19
Keywords: oral antivirals; high risk patients
MeSH Terms: conditions — COVID-19 | interventions — Antiviral Agents; nirmatrelvir and ritonavir drug combination; molnupiravir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Oral Antiviral Group: Study participant initiated with oral antiviral (nirmatrelvir plus ritonavir or molnupiravir) for the treatment of COVID-19
  Interventions: Drug: Oral Antiviral
- Non Oral Antiviral Group: Study participant not initiated with oral antiviral for the treatment of COVID-19

INTERVENTIONS:
Drug: Oral Antiviral — Nirmatrelvir plus ritonavir or molnupiravir
  Other Names: Paxlovid; Lagevrio
  Groups: Oral Antiviral Group

SUMMARY:
This study is a prospective observational cohort study to evaluate the benefit of oral antivirals (nirmatrelvir plus ritonavir or molnupiravir) in Ministry of Health institutions. In this study, we will observe the progress of COVID-19 study participants seen in the health clinic up to 90 days from their initial visit to the health clinic.

DETAILED DESCRIPTION:
This protocol is a prospective, multi-center, observational cohort study to evaluate the benefit of oral antivirals (nirmatrelvir plus ritonavir or molnupiravir) in Ministry of Health institutions in preventing progression of COVID-19 to severe COVID-19.

In this study, we will observe the clinical outcomes (COVID-19 symptoms, hospitalization admission, mortality, long term COVID-19 symptoms) of COVID-19 study participants seen in the health clinic up to 90 days from their initial visit to the health clinic . The hypothesis is that oral antiviral is beneficial in preventing disease progression and reducing long term COVID-19 symptoms.

ELIGIBILITY:
Inclusion Criteria:

* All SARS-CoV-2 positive individuals who are eligible for oral antiviral treatment based on current Ministry of Health Malaysia guidelines.

Exclusion Criteria:

* Individual who received oral antiviral (either nirmatrelvir plus ritonavir or monupiravir) more than 5 days following their positive SARS-CoV-2 test date

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All SARS-CoV-2 positive adult population seen in the Ministry of Health Malaysia institutions
Sampling Method: Non-Probability Sample
Enrollment: 660 (Estimated)
Dates: Start 2022-12-06 (Actual); Primary Completion 2023-07-30 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Frequency and proportion of study participants with COVID-19 related Hospitalization | Within 28 days after treatment initiation
  Hospital admission due to COVID-19
Frequency and proportion of of study participants with COVID-19 related all-caused mortality | Within 28 days after treatment initiation
  Any cause of death

SECONDARY OUTCOMES:
Frequency and proportion of study participants with of COVID-19 related symptoms | Within 28 days after treatment initiation
  Type of COVID-19 related symptoms (Eg. fever or chills, fatigue, shortness of breath, new loss of taste or smell, sore throat, congestion or runny nose, nausea or vomiting, diarrhea)
Frequency and proportion of study participants with COVID-19 ICU admission | Within 28 days after treatment initiation
  Admission to Intensive Care Unit (ICU) due to COVID-19
Frequency and proportion of study participants with adverse drug reaction | Within 28 days after treatment initiation
  Medication related adverse reaction (eg. rash, itchiness, increased blood pressure, abdominal pain, etc)
Duration of Hospitalization | Within 28 days after treatment initiation
  Number of days hospitalized due to COVID-19
Frequency and proportion of study participants with long-term COVID-19 symptoms | COVID-19 related symptoms lasting more than 4 weeks up to 6 months following COVID-19
  COVID-19 related symptoms that last more than 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ee Vien Low, Ph.D., Principal Investigator — Clinical Research Center, Malaysia
Locations (8):
- Malaysia (8):
  - Klinik Kesihatan Kajang, Kajang, Selangor
  - Klinik Kesihatan Banadar Botanik, Klang, Selangor
  - Klinik Kesihatan Bukit Kuda, Klang, Selangor
  - Klinik Kesihatan Pandamaran, Klang, Selangor
  - Klinik Kesihatan Seksyen 19, Petaling Jaya, Selangor
  - Klinik Kesihatan Seksyen 7, Petaling Jaya, Selangor
  - Klinik Kesihatan Puchong Batu 14, Subang Jaya, Selangor
  - Klinik Kesihatan Taman Medan, Petaling Jaya